CLINICAL TRIAL: NCT03941964
Title: A Phase 3b, Single-Arm, Multicenter Open-Label Study of Venetoclax in Combination With Azacitidine or Decitabine in an Outpatient Setting in AML Patients Ineligible for Intensive Chemotherapy
Brief Title: A Study of the Effectiveness of Venetoclax in Combination With Azacitidine or Decitabine in an Outpatient Setting in Patients With Acute Myeloid Leukemia (AML) Ineligible for Intensive Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M19-072
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2019-05-03; First posted 2019-05-08 (Actual); Results first posted 2023-03-20 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-02

CONDITIONS: Acute Myeloid Leukemia (AML); Cancer
Keywords: Acute Myeloid Leukemia (AML); Cancer; Treatment-naïve; Venetoclax; Azacitidine; Decitabine; Outpatient setting
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — venetoclax; Azacitidine; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Venetoclax 400 mg + azacitidine 75 mg (Experimental): Participants received venetoclax orally daily for 28-day cycles, for a maximum of 6 cycles, beginning on Cycle 1 Day 1. The venetoclax dosing ramp-up schedule was 100 mg on Cycle 1 Day 1, 200 mg on Cycle 1 Day 2, and 400 mg on Cycle 1 Days 3 -28 and 400 mg daily for each 28-day cycle thereafter. Azacitidine (75 mg/m^2) was administered subcutaneously or intravenously per investigator's choice and institutional practice for 7 days beginning on Day 1 of each 28-day cycle.
  Interventions: Drug: Venetoclax; Drug: Azacitidine
- Venetoclax 400 mg + decitabine 20 mg (Experimental): Participants received venetoclax orally daily for 28-day cycles, for a maximum of 6 cycles, beginning on Cycle 1 Day 1. The venetoclax dosing ramp-up schedule was 100 mg on Cycle 1 Day 1, 200 mg on Cycle 1 Day 2, and 400 mg on Cycle 1 Days 3 -28 and 400 mg daily for each 28-day cycle thereafter. Decitabine (20 mg/m^2) was administered intravenously per investigator's choice and institutional practice for 5 days beginning on Day 1 of each cycle.
  Interventions: Drug: Venetoclax; Drug: Decitabine

INTERVENTIONS:
Drug: Venetoclax — Venetoclax tablets were to be taken orally once daily with a meal and water in the morning at approximately the same time each day. Tablets were to be swallowed whole and not chewed, crushed, or broken prior to swallowing. On the days that the participant received either azacitidine or decitabine, venetoclax was dosed in clinic and administered prior to these agents.
  Other Names: ABT-199; VENCLEXTA; VENCLYXTO
Drug: Azacitidine — The azacitidine infusion was prepared and administered per the package insert and given either subcutaneously or intravenously, per institutional practice.
  Other Names: Vidaza
  Arms: Venetoclax 400 mg + azacitidine 75 mg
Drug: Decitabine — The decitabine infusion was prepared and administered per the package insert and given intravenously, per institutional practice.
  Other Names: Dacogen
  Arms: Venetoclax 400 mg + decitabine 20 mg

SUMMARY:
A study evaluating the effectiveness and safety of venetoclax, in combination with azacitidine or decitabine, in an outpatient setting for treatment-naïve participants with AML who are ineligible for intensive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant has confirmation of acute myeloid leukemia (AML) by World Health Organization (WHO) criteria
* Participant is deemed by the investigator to be an appropriate candidate for outpatient ramp-up of venetoclax
* Participant is not eligible to receive treatment with standard cytarabine and anthracycline induction regimens
* Participant has not received prior treatment for AML (treatment naïve) with the exception of hydroxyurea
* Participant has no evidence of spontaneous tumor lysis syndrome (TLS) at Screening
* Participant can have progressed from myelodysplastic syndrome (MDS) or be considered to have secondary AML and could have been treated with growth factors or other agents with the exception of hypomethylating agents
* Participant has adequate kidney, liver, and hematology laboratory values as detailed in the protocol
* Has an Eastern Cooperative Oncology Group (ECOG) Performance status of 0 to 3

Exclusion Criteria:

Has a history of the following conditions:

* Acute promyelocytic leukemia
* Known active central nervous system involvement with AML
* Positive for HIV (HIV testing is not required)
* Positive for hepatitis B or C infection with the exception of those with an undetectable viral load within 3 months
* Cardiovascular disability status of New York Heart Association Class > 2
* Chronic respiratory disease that requires continuous oxygen or any other medical condition that in the opinion of the investigator would adversely affect his/her participating in this study
* Malabsorption syndrome or other condition that precludes enteral route of administration

Has a history of other malignancies within 2 years prior to study entry, with the exception of:

* Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast
* Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin
* Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (16):
- United States (16):
  - Arizona Oncology Associates, PC-HOPE /ID# 211509, Tempe, Arizona
  - Colorado Blood Cancer Institute /ID# 212800, Denver, Colorado
  - Rocky Mountain Cancer Centers /ID# 211508, Lone Tree, Colorado
  - Fort Wayne Medical Oncology /ID# 223523, Fort Wayne, Indiana
  - Minnesota Oncology Hematology, PA /ID# 212837, Minneapolis, Minnesota
  - Oncology Hematology Care, Inc. /ID# 212779, Cincinnati, Ohio
  - Willamette Valley Cancer Institute and Research Center /ID# 211504, Eugene, Oregon
  - Charleston Oncology, P.A. /ID# 211471, Charleston, South Carolina
  - Prisma Health Cancer Inst - Eastside /ID# 211466, Greenville, South Carolina
  - Tennessee Oncology - Chattanooga / McCallie /ID# 212717, Chattanooga, Tennessee
  - Tennessee Oncology-Nashville Centennial /ID# 210944, Nashville, Tennessee
  - Texas Oncology - Austin Midtown /ID# 212780, Austin, Texas
  - Texas Oncology - Medical City Dallas /ID# 211503, Dallas, Texas
  - Texas Transplant Institute /ID# 213311, San Antonio, Texas
  - Texas Oncology - San Antonio Medical Center /ID# 211510, San Antonio, Texas
  - Texas Oncology - Northeast Texas /ID# 213908, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Manda S, Anz BM 3rd, Benton C, Broun ER, Yimer HA, Renshaw JS, Geils G Jr, Berdeja J, Cruz J, Melear JM, Fanning S, Fletcher L, Li Y, Duan Y, Werner ME, Potluri J, Pai MV, Donnellan WB. A phase 3b study of venetoclax and azacitidine or decitabine in an outpatient setting in patients with acute myeloid leukemia. Hematol Oncol. 2024 May;42(3):e3274. doi: 10.1002/hon.3274. PMID 38711253
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants who received at least one dose of venetoclax and azacitidine or decitabine; this study disposition represents the primary reason for venetoclax discontinuation
Period: Overall Study
Arm/Group | Venetoclax 400 mg + Azacitidine 75 mg | Venetoclax 400 mg + Decitabine 20 mg
Started | 30 | 30
Completed | 7 | 11
Not Completed | 23 | 19
Not completed — Adverse Event | 1 | 8
Not completed — Progressive disease | 7 | 3
Not completed — Lack of Efficacy | 0 | 1
Not completed — Death | 3 | 1
Not completed — Withdrew consent | 1 | 3
Not completed — Physician Decision | 9 | 2
Not completed — Other, not specified | 2 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of venetoclax and azacitidine or decitabine
Groups:
- Total: Total of all reporting groups
Arm/Group | Venetoclax 400 mg + Azacitidine 75 mg | Venetoclax 400 mg + Decitabine 20 mg | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.0 (6.31) | 76.2 (6.35) | 76.6 (6.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 15 | 14 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 26 | 29 | 55
  Black or African American | 4 | 1 | 5
  Asian | 0 | 0 | 0
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Remission or Complete Remission With Incomplete Blood Count Recovery (CR + CRi)
Description: The composite complete remission rate is defined as the percentage of participants with complete remission (CR) or complete remission with incomplete blood count recovery (CRi) at any time during the study as assessed by the investigator. Response was based on bone marrow results and hematology values according to the modified International Working Group (IWG) criteria for AML:
  CR: Absolute neutrophil count (ANC) > 10^3/μL (1,000/μL), platelets > 10^5/μL (100,000/μL), red blood cell (RBC) transfusion independence, and bone marrow with < 5% blasts
  CRi: Bone marrow with < 5% blasts, and absolute neutrophils of ≤ 10^3/μL or platelets ≤ 10^5/μL
Time Frame: Assessed at Cycle 1 end, at Cycle 2 end if CR/CRi wasn't achieved at Cycle 1 end, or Cycle 4 end if CR/CRi wasn't achieved at Cycle 2 end. Median treatment duration of venetoclax was 16.1 wks (range 3.9-38.1) and 21.1 wks (range 2.7-40.4), respectively.
Population: All participants who received at least one dose of venetoclax and azacitidine or decitabine
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax 400 mg + Azacitidine 75 mg | Venetoclax 400 mg + Decitabine 20 mg
Number analyzed (Participants) | 30 | 30
percentage of participants | 70.0 [50.6 to 85.3] | 63.3 [43.9 to 80.1]

2. Secondary Outcome: Percentage of Participants With Complete Remission (CR)
Description: The complete remission rate is defined as the percentage of participants with complete remission (CR) at any time during the study as assessed by the investigator. Response was based on bone marrow results and hematology values according to the modified International Working Group (IWG) criteria for AML:
  CR: Absolute neutrophil count (ANC) > 10^3/μL (1,000/μL), platelets > 10^5/μL (100,000/μL), red blood cell (RBC) transfusion independence, and bone marrow with < 5% blasts
Time Frame: as for outcome 1
Population: All participants who received at least one dose of venetoclax and azacitidine or decitabine
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax 400 mg + Azacitidine 75 mg | Venetoclax 400 mg + Decitabine 20 mg
Number analyzed (Participants) | 30 | 30
percentage of participants | 13.3 [3.8 to 30.7] | 26.7 [12.3 to 45.9]

3. Secondary Outcome: Percentage of Participants With Complete Remission With Incomplete Blood Count Recovery (CRi)
Description: The complete remission with incomplete blood count recovery rate is defined as the percentage of participants with complete remission with incomplete blood count recovery (CRi) at any time during the study as assessed by the investigator. Response was based on bone marrow results and hematology values according to the modified International Working Group (IWG) criteria for AML:
  CRi: Bone marrow with < 5% blasts, and absolute neutrophils of ≤ 10^3/μL or platelets ≤ 10^5/μL.
Time Frame: as for outcome 1
Population: All participants who received at least one dose of venetoclax and azacitidine or decitabine
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax 400 mg + Azacitidine 75 mg | Venetoclax 400 mg + Decitabine 20 mg
Number analyzed (Participants) | 30 | 30
percentage of participants | 56.7 [37.4 to 74.5] | 36.7 [19.9 to 56.1]

4. Secondary Outcome: Percentage of Participants With Post-baseline Transfusion Independence
Description: The transfusion independence rate is defined as the percentage of participants with post-baseline transfusion independence, which is defined as a period of at least 56 days with no transfusion after the first dose of study drug and within 30 days of the last dose of study drug, death, or initiation of post-treatment therapy, whichever is earliest.
Time Frame: From the first dose of study drug to the last dose of study drug +30 days, or death, or initiation of post-treatment therapy, whichever occurred earliest. Median time on follow-up was 183.5 days and 195.0 days, respectively.
Population: All participants who received at least one dose of venetoclax and azacitidine or decitabine
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Venetoclax 400 mg + Azacitidine 75 mg | Venetoclax 400 mg + Decitabine 20 mg
Number analyzed (Participants) | 30 | 30
percentage of participants
  Red blood cells (RBC) | 50.0 [31.3 to 68.7] | 60.0 [40.6 to 77.3]
  Platelets | 73.3 [54.1 to 87.7] | 73.3 [54.1 to 87.7]
  RBC and platelets | 50.0 [31.3 to 68.7] | 60.0 [40.6 to 77.3]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to end of study; median time on follow up was 183.5, 195.0 and 195.0 days, respectively. TEAEs and SAEs were collected from first dose of study drug until 30 days after last dose of study drug; mean time on venetoclax was 18.2, 18.6, and 18.4 weeks, respectively.
Groups:
- Venetoclax 400 mg + Azacitidine 75 mg or Decitabine 20 mg: Participants received venetoclax orally daily for 28-day cycles, for a maximum of 6 cycles, beginning on Cycle 1 Day 1. The venetoclax dosing ramp-up schedule was 100 mg on Cycle 1 Day 1, 200 mg on Cycle 1 Day 2, and 400 mg on Cycle 1 Days 3 -28 and 400 mg daily for each 28-day cycle thereafter. Azacitidine (75 mg/m^2) was administered subcutaneously or intravenously per investigator's choice and institutional practice for 7 days beginning on Day 1 of each 28-day cycle. Decitabine (20 mg/m^2) was administered intravenously per investigator's choice and institutional practice for 5 days beginning on Day 1 of each cycle.
Arm/Group | Venetoclax 400 mg + Azacitidine 75 mg | Venetoclax 400 mg + Decitabine 20 mg | Venetoclax 400 mg + Azacitidine 75 mg or Decitabine 20 mg
All-Cause Mortality (participants affected / at risk) | 5/30 | 8/30 | 13/60
Serious Adverse Events (participants affected / at risk) | 19/30 | 22/30 | 41/60
Other Adverse Events (participants affected / at risk) | 29/30 | 30/30 | 59/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax 400 mg + Azacitidine 75 mg (N=30) | Venetoclax 400 mg + Decitabine 20 mg (N=30) | Venetoclax 400 mg + Azacitidine 75 mg or Decitabine 20 mg (N=60)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 8 (11) | 10 (12) | 18 (23)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (4) | 1 (4)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (6) | 1 (6)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 (3) | 1 (1) | 3 (4)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
PROCTALGIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 1 (1)
DEATH (General disorders) | 2 (2) | 2 (2) | 4 (4)
DISEASE PROGRESSION (General disorders) | 2 (2) | 1 (1) | 3 (3)
PYREXIA (General disorders) | 0 (0) | 3 (3) | 3 (3)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PERINEAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
SEPSIS (Infections and infestations) | 2 (3) | 8 (10) | 10 (13)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 3 (3) | 0 (0) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Venetoclax 400 mg + Azacitidine 75 mg (N=30) | Venetoclax 400 mg + Decitabine 20 mg (N=30) | Venetoclax 400 mg + Azacitidine 75 mg or Decitabine 20 mg (N=60)
ANAEMIA (Blood and lymphatic system disorders) | 23 (46) | 24 (79) | 47 (125)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
NEUTROPENIA (Blood and lymphatic system disorders) | 3 (5) | 9 (18) | 12 (23)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 3 (4) | 10 (23) | 13 (27)
ATRIAL FIBRILLATION (Cardiac disorders) | 3 (3) | 1 (1) | 4 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 6 (7) | 8 (9)
CONSTIPATION (Gastrointestinal disorders) | 11 (15) | 8 (10) | 19 (25)
DIARRHOEA (Gastrointestinal disorders) | 12 (15) | 11 (15) | 23 (30)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 3 (3) | 4 (5) | 7 (8)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 17 (23) | 15 (22) | 32 (45)
STOMATITIS (Gastrointestinal disorders) | 3 (3) | 4 (7) | 7 (10)
VOMITING (Gastrointestinal disorders) | 13 (15) | 3 (4) | 16 (19)
CHEST PAIN (General disorders) | 0 (0) | 2 (3) | 2 (3)
CHILLS (General disorders) | 0 (0) | 4 (4) | 4 (4)
FATIGUE (General disorders) | 13 (14) | 12 (18) | 25 (32)
INJECTION SITE REACTION (General disorders) | 3 (3) | 0 (0) | 3 (3)
MALAISE (General disorders) | 2 (2) | 0 (0) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 8 (10) | 7 (8) | 15 (18)
PYREXIA (General disorders) | 6 (8) | 7 (8) | 13 (16)
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
FUNGAL SKIN INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
PNEUMONIA (Infections and infestations) | 2 (2) | 2 (2) | 4 (4)
SINUSITIS (Infections and infestations) | 1 (1) | 2 (3) | 3 (4)
URINARY TRACT INFECTION (Infections and infestations) | 4 (5) | 1 (1) | 5 (6)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 4 (4)
FALL (Injury, poisoning and procedural complications) | 5 (6) | 5 (6) | 10 (12)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 2 (3) | 4 (5)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 2 (5) | 4 (7)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (4) | 4 (5) | 7 (9)
BLOOD CREATININE INCREASED (Investigations) | 2 (2) | 1 (3) | 3 (5)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (3) | 4 (46) | 6 (49)
NEUTROPHIL COUNT DECREASED (Investigations) | 19 (54) | 15 (92) | 34 (146)
PLATELET COUNT DECREASED (Investigations) | 14 (54) | 16 (80) | 30 (134)
WEIGHT DECREASED (Investigations) | 8 (13) | 1 (1) | 9 (14)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 15 (45) | 16 (114) | 31 (159)
DECREASED APPETITE (Metabolism and nutrition disorders) | 10 (10) | 2 (2) | 12 (12)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 5 (5)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (3) | 2 (2) | 3 (5)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 4 (5)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 3 (3) | 7 (11) | 10 (14)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 1 (2) | 2 (2) | 3 (4)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 (2) | 3 (6) | 5 (8)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5) | 7 (7)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 8 (8)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 3 (5)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 3 (4)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 7 (7)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 5 (5)
DIZZINESS (Nervous system disorders) | 3 (3) | 5 (6) | 8 (9)
HEADACHE (Nervous system disorders) | 4 (5) | 4 (5) | 8 (10)
PRESYNCOPE (Nervous system disorders) | 2 (3) | 0 (0) | 2 (3)
ANXIETY (Psychiatric disorders) | 3 (3) | 0 (0) | 3 (3)
CONFUSIONAL STATE (Psychiatric disorders) | 2 (2) | 1 (1) | 3 (3)
DEPRESSION (Psychiatric disorders) | 2 (2) | 3 (3) | 5 (5)
INSOMNIA (Psychiatric disorders) | 5 (6) | 6 (7) | 11 (13)
DYSURIA (Renal and urinary disorders) | 0 (0) | 2 (4) | 2 (4)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5) | 11 (11)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4) | 4 (5)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5) | 4 (6)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 4 (4)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5) | 5 (7)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 4 (4)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (4) | 5 (7)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)
HYPOTENSION (Vascular disorders) | 3 (3) | 4 (5) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/64/NCT03941964/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/64/NCT03941964/SAP_001.pdf